CLINICAL TRIAL: NCT03789318
Title: A Phase 2, Randomized, Double-blind, Placebo-Controlled Efficacy, Pharmacokinetics and Safety Study of CA-008 in Subjects Undergoing Complete Abdominoplasty
Brief Title: Study in Subjects Undergoing Complete Abdominoplasty
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Concentric Analgesics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CA-PS-204
Record Dates: First submitted 2018-12-02; First posted 2018-12-28 (Actual); Results first posted 2022-01-13 (Actual); Last update posted 2024-03-19 (Actual); Status verified 2024-03

CONDITIONS: Postsurgical Pain
MeSH Terms: conditions — Pain, Postoperative | interventions — Bupivacaine; Hydromorphone; Fentanyl; Acetaminophen; Oxycodone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- CA-008 5 mg (0.05 mg/mL) Cohort 1 (Active Comparator): Cohort 1 (CA-008 5 mg): the surgery for each subject is to be performed under general anesthesia supplemented by a transverse abdominis plane (TAP) block and local surgical site infiltration. Prior to the surgery, perform the TAP block as a single injection of 0.25% bupivacaine hydrochloride (HCl) 60 mL (150 mg).
  Interventions: Drug: CA-008 5 mg; Drug: Bupivacaine Hydrochloride; Drug: Hydromorphone; Drug: Fentanyl; Drug: Acetaminophen; Drug: Oxycodone
- Placebo for Cohort 1 (Placebo Comparator): Cohort 1:
  Placebo comparator is identical in appearance to the investigational product, containing the same excipients as the active comparator.
  The surgery for each subject is to be performed under general anesthesia supplemented by a transverse abdominis plane (TAP) block and local surgical site infiltration. Prior to the surgery, perform the TAP block as a single injection of 0.25% bupivacaine hydrochloride (HCl) 60 mL (150 mg).
  Interventions: Drug: Placebo; Drug: Bupivacaine Hydrochloride; Drug: Hydromorphone; Drug: Fentanyl; Drug: Acetaminophen; Drug: Oxycodone
- CA-008 10 mg (0.1 mg/mL) (Active Comparator): Cohort 2 (CA-008 10 mg): the surgery is to be performed under general anesthesia supplemented by a transverse abdominis plane (TAP) block and local surgical site infiltration. Prior to the surgery, perform the TAP block as a single injection of 0.25% bupivacaine hydrochloride (HCl) 60 mL (150 mg).
  Interventions: Drug: Bupivacaine Hydrochloride; Drug: Hydromorphone; Drug: Fentanyl; Drug: Acetaminophen; Drug: Oxycodone; Drug: CA-008 10 mg
- CA-008 15 mg (0.15 mg/mL) (Active Comparator): Cohort 3 (CA-008 15 mg): the surgery is to be performed under general anesthesia supplemented by a transverse abdominis plane (TAP) block and local surgical site infiltration. Prior to the surgery, perform the TAP block as a single injection of 0.25% bupivacaine hydrochloride (HCl) 60 mL (150 mg).
  Interventions: Drug: Bupivacaine Hydrochloride; Drug: Hydromorphone; Drug: Fentanyl; Drug: Acetaminophen; Drug: Oxycodone; Drug: CA-008 15 mg
- Placebo for Cohorts 2 and 3 (Placebo Comparator): Cohorts 2 & 3:
  Placebo comparator in each cohort is identical in appearance to the investigational product, containing the same excipients as the active comparator.
  The surgery for each subject is to be performed under general anesthesia supplemented by a transverse abdominis plane (TAP) block and local surgical site infiltration. Prior to the surgery, perform the TAP block as a single injection of 0.25% bupivacaine hydrochloride (HCl) 60 mL (150 mg).
  Interventions: Drug: Placebo; Drug: Bupivacaine Hydrochloride; Drug: Hydromorphone; Drug: Fentanyl; Drug: Acetaminophen; Drug: Oxycodone

INTERVENTIONS:
Drug: CA-008 5 mg — 5 mg CA-008 reconstituted in saline.
  Other Names: Vocacapsaicin
  Arms: CA-008 5 mg (0.05 mg/mL) Cohort 1
Drug: Placebo — Each cohort will use placebo reconstituted in saline.
  Arms: Placebo for Cohort 1; Placebo for Cohorts 2 and 3
Drug: Bupivacaine Hydrochloride — 0.25% administered pre-surgery
Drug: Hydromorphone — 0.02 mg/kg IV administered intraoperatively
Drug: Fentanyl — 100 mcg IV administered intraoperatively
Drug: Acetaminophen — 1000 mg IV administered intraoperatively
Drug: Oxycodone — 5-10 mg PO administered post-surgery
Drug: CA-008 10 mg — 10 mg CA-008 reconstituted in saline.
  Other Names: Vocacapsaicin
  Arms: CA-008 10 mg (0.1 mg/mL)
Drug: CA-008 15 mg — 15 mg CA-008 reconstituted in saline.
  Other Names: Vocacapsaicin
  Arms: CA-008 15 mg (0.15 mg/mL)

SUMMARY:
Phase 2, single center, randomized, double-blind, placebo-controlled, parallel design study of CA-008 vs. placebo in subjects undergoing an elective C-ABD under general anesthesia supplemented with a bupivacaine hydrochloride (HCl)transverse abdominis plane (TAP) block.

DETAILED DESCRIPTION:
This is a Phase 2, single-center, randomized, double-blind, placebo-controlled, parallel design study evaluating up to 4 ascending dose level cohorts, each evaluating a single dose of CA-008 vs. placebo injected/instilled during an elective C-ABD. Up to 72 subjects may be randomized in 4 cohorts.

For each subject, postsurgical assessments will be conducted in two parts:

* Inpatient period: starts with completion of study treatment injection (T0) and continues through 96 hours (T96h).
* Outpatient period: begins on discharge from the inpatient unit through various follow up visits to day 29 (D29)/week 4 (W4) after surgery. Note that additional follow up visits may occur at any time or even after D29/W4 to follow adverse events (AEs) to resolution or establishment of a new baseline.

ELIGIBILITY:
Key Inclusion Criteria:

* Plan to undergo an elective complete abdominoplasty (C-ABD), without collateral procedure or additional surgeries.
* In the medical judgment of the investigator, be a reasonably healthy adult aged 18 - 65 years old, inclusive, and American Society of Anesthesiology (ASA) physical Class 1 or 2 at the time of randomization.
* Unless the subject has a same sex partner, he or she must either be sterile (surgically or biologically) or commit to an acceptable method of birth control while participating in the study.
* Have a body mass index ≤ 35 kg/m².
* Be willing and able to sign the informed consent form (ICF) approved by an Institutional Review Board (IRB).

Key Exclusion Criteria:

* In the opinion of the Investigator, have a concurrent painful condition that may require analgesic treatment during the study period or may confound post-surgical pain assessments.
* Have a known allergy to chili peppers, capsaicin or the components of CA-008, acetaminophen, bupivacaine, fentanyl hydromorphone or oxycodone.
* As determined by the investigator have a history or clinical manifestation of significant medical, neuropsychiatric or other condition, including a clinically significant existing arrhythmia, left bundle branch block or abnormal ECG, myocardial infarction or coronary arterial bypass graft surgery within the prior 12 months, significant abnormal clinical laboratory test value, or known bleeding abnormality that could preclude or impair study participation or interfere with study assessments.
* The following are considered disallowed medications:

  1. Be tolerant to opioids defined as those who have been receiving or have received chronic opioid therapy greater than 15 mg of oral morphine equivalents per day for greater than 3 out of 7 days per week over a one-month period within 6 months of screening.
  2. Within 1 day prior to surgery and throughout the inpatient period, be taking any capsaicin-containing products, such as dietary supplements or over-the-counter (OTC) preparations, including topical formulations, and prescription medications.
  3. Within the 7 days prior to surgery, be taking any central nervous system (CNS) active agent as an analgesic adjunct medication, such as anticonvulsants, antidepressants, benzodiazepines, sedative- hypnotics, clonidine and other central alpha-2 agents, ketamine or muscle relaxants.

  i. These drugs are permitted if prescribed for non-pain indications and the dose has been stable for at least 30 days prior to surgery.

ii. The use of benzodiazepines and the non-benzodiazepines are permitted to treat insomnia during the postoperative period.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2018-12-03 (Actual); Primary Completion 2019-05-16 (Actual); Study Completion 2019-06-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Alina Beaton, MD, Principal Investigator — Lotus Clinical Research, LLC
Locations (1):
- Lotus Clinical Research, LLC, Pasadena, California, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo for Cohort 1: Cohort 1: the surgery for each subject is to be performed under general anesthesia supplemented by a transverse abdominis plane (TAP) block and local surgical site infiltration. Prior to the surgery, perform the TAP block as a single injection of 0.25% bupivacaine hydrochloride (HCl) 60 mL (150 mg).
  Placebo: Each cohort will use placebo reconstituted in saline.
  Bupivacaine Hydrochloride: 0.25% administered pre-surgery
  Hydromorphone: 0.02 mg/kg IV administered intraoperatively
  Fentanyl: 100 mcg IV administered intraoperatively
  Acetaminophen: 1000 mg IV administered intraoperatively
  Oxycodone: 5-10 mg PO administered post-surgery
- CA-008 10 mg (0.1 mg/mL) Cohort 2: Cohort 2 (CA-008 10 mg): the surgery is to be performed under general anesthesia supplemented by a transverse abdominis plane (TAP) block and local surgical site infiltration. Prior to the surgery, perform the TAP block as a single injection of 0.25% bupivacaine hydrochloride (HCl) 60 mL (150 mg).
  Bupivacaine Hydrochloride: 0.25% administered pre-surgery
  Hydromorphone: 0.02 mg/kg IV administered intraoperatively
  Fentanyl: 100 mcg IV administered intraoperatively
  Acetaminophen: 1000 mg IV administered intraoperatively
  Oxycodone: 5-10 mg PO administered post-surgery
  CA-008 10 mg: 10 mg CA-008 reconstituted in saline.
- CA-008 15 mg (0.15 mg/mL) Cohort 3: Cohort 3 (CA-008 15 mg): the surgery is to be performed under general anesthesia supplemented by a transverse abdominis plane (TAP) block and local surgical site infiltration. Prior to the surgery, perform the TAP block as a single injection of 0.25% bupivacaine hydrochloride (HCl) 60 mL (150 mg).
  Bupivacaine Hydrochloride: 0.25% administered pre-surgery
  Hydromorphone: 0.02 mg/kg IV administered intraoperatively
  Fentanyl: 100 mcg IV administered intraoperatively
  Acetaminophen: 1000 mg IV administered intraoperatively
  Oxycodone: 5-10 mg PO administered post-surgery
  CA-008 15 mg: 15 mg CA-008 reconstituted in saline.
- Placebo for Cohorts 2 and 3: Cohorts 2 & 3: the surgery for each subject is to be performed under general anesthesia supplemented by a transverse abdominis plane (TAP) block and local surgical site infiltration. Prior to the surgery, perform the TAP block as a single injection of 0.25% bupivacaine hydrochloride (HCl) 60 mL (150 mg).
  Placebo: Each cohort will use placebo reconstituted in saline.
  Bupivacaine Hydrochloride: 0.25% administered pre-surgery
  Hydromorphone: 0.02 mg/kg IV administered intraoperatively
  Fentanyl: 100 mcg IV administered intraoperatively
  Acetaminophen: 1000 mg IV administered intraoperatively
  Oxycodone: 5-10 mg PO administered post-surgery
Period: Overall Study
Arm/Group | CA-008 5 mg (0.05 mg/mL) Cohort 1 | Placebo for Cohort 1 | CA-008 10 mg (0.1 mg/mL) Cohort 2 | CA-008 15 mg (0.15 mg/mL) Cohort 3 | Placebo for Cohorts 2 and 3
Started | 9 | 9 | 12 | 12 | 12
Completed | 9 | 9 | 9 | 11 | 12
Not Completed | 0 | 0 | 3 | 1 | 0
Not completed — Adverse Event | 0 | 0 | 1 | 1 | 0
Not completed — Lost to Follow-up | 0 | 0 | 1 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- CA-008 5 mg (0.05 mg/mL) Cohort 1: Cohort 1 (CA-008 5 mg): the surgery for each subject is to be performed under general anesthesia supplemented by a transverse abdominis plane (TAP) block and local surgical site infiltration. Prior to the surgery, perform the TAP block as a single injection of 0.25% bupivacaine hydrochloride (HCl) 60 mL (150 mg).
  CA-008 5 mg: 5 mg CA-008
  Bupivacaine Hydrochloride: 0.25% administered pre-surgery
  Hydromorphone: 0.02 mg/kg IV administered intraoperatively
  Fentanyl: 100 mcg IV administered intraoperatively
  Acetaminophen: 1000 mg IV administered intraoperatively
  Oxycodone: 5-10 mg PO administered post-surgery
- Placebo for Cohort 1: Cohort 1:
  Placebo comparator is identical in appearance to the investigational product, containing the same excipients as the active.
  The surgery for each subject is to be performed under general anesthesia supplemented by a transverse abdominis plane (TAP) block and local surgical site infiltration. Prior to the surgery, perform the TAP block as a single injection of 0.25% bupivacaine hydrochloride (HCl) 60 mL (150 mg).
  Placebo: Each cohort will use placebo reconstituted in saline.
  Bupivacaine Hydrochloride: 0.25% administered pre-surgery
  Hydromorphone: 0.02 mg/kg IV administered intraoperatively
  Fentanyl: 100 mcg IV administered intraoperatively
  Acetaminophen: 1000 mg IV administered intraoperatively
  Oxycodone: 5-10 mg PO administered post-surgery
- CA-008 10 mg (0.1 mg/mL): Cohort 2 (CA-008 10 mg): the surgery is to be performed under general anesthesia supplemented by a transverse abdominis plane (TAP) block and local surgical site infiltration. Prior to the surgery, perform the TAP block as a single injection of 0.25% bupivacaine hydrochloride (HCl) 60 mL (150 mg).
  Bupivacaine Hydrochloride: 0.25% administered pre-surgery
  Hydromorphone: 0.02 mg/kg IV administered intraoperatively
  Fentanyl: 100 mcg IV administered intraoperatively
  Acetaminophen: 1000 mg IV administered intraoperatively
  Oxycodone: 5-10 mg PO administered post-surgery
  CA-008 10 mg: 10 mg CA-008
- CA-008 15 mg (0.15 mg/mL): Cohort 3 (CA-008 15 mg): the surgery is to be performed under general anesthesia supplemented by a transverse abdominis plane (TAP) block and local surgical site infiltration. Prior to the surgery, perform the TAP block as a single injection of 0.25% bupivacaine hydrochloride (HCl) 60 mL (150 mg).
  Bupivacaine Hydrochloride: 0.25% administered pre-surgery
  Hydromorphone: 0.02 mg/kg IV administered intraoperatively
  Fentanyl: 100 mcg IV administered intraoperatively
  Acetaminophen: 1000 mg IV administered intraoperatively
  Oxycodone: 5-10 mg PO administered post-surgery
  CA-008 15 mg: 15 mg CA-008
- Placebo for Cohorts 2 and 3: Cohorts 2 & 3:
  Placebo comparator in each cohort is identical in appearance to the investigational product, containing the same excipients as the active.
  The surgery for each subject is to be performed under general anesthesia supplemented by a transverse abdominis plane (TAP) block and local surgical site infiltration. Prior to the surgery, perform the TAP block as a single injection of 0.25% bupivacaine hydrochloride (HCl) 60 mL (150 mg).
  Placebo: Each cohort will use placebo reconstituted in saline.
  Bupivacaine Hydrochloride: 0.25% administered pre-surgery
  Hydromorphone: 0.02 mg/kg IV administered intraoperatively
  Fentanyl: 100 mcg IV administered intraoperatively
  Acetaminophen: 1000 mg IV administered intraoperatively
  Oxycodone: 5-10 mg PO administered post-surgery
- Total: Total of all reporting groups
Arm/Group | CA-008 5 mg (0.05 mg/mL) Cohort 1 | Placebo for Cohort 1 | CA-008 10 mg (0.1 mg/mL) | CA-008 15 mg (0.15 mg/mL) | Placebo for Cohorts 2 and 3 | Total
Number analyzed (Participants) | 9 | 9 | 12 | 12 | 12 | 54
Age, Continuous [Mean (Standard Deviation); unit: years] | 37.8 (10.95) | 38.2 (7.17) | 43.3 (10.27) | 43.3 (6.74) | 38.3 (8.76) | 40.4 (8.93)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 9 | 12 | 12 | 12 | 54
  Male | 0 | 0 | 0 | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 5 | 6 | 4 | 6 | 4 | 25
  Not Hispanic or Latino | 4 | 3 | 8 | 6 | 8 | 29
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 1 | 0 | 1 | 1 | 0 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 1 | 1
  Black or African American | 1 | 1 | 6 | 3 | 6 | 17
  White | 7 | 8 | 5 | 8 | 5 | 33
  More than one race | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 9 | 9 | 12 | 12 | 12 | 54

OUTCOME MEASURES:

1. Primary Outcome: Pain Intensity Scores at 96 Hours at Rest Using Numerical Rating Scale (NRS)
Description: Numeric Rating Scale (NRS) of pain intensity from 0-10 where 0 is no pain and 10 is the worst pain imaginable at 96 hours
Time Frame: 96 hours
Population: Safety population
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Placebo for Cohort 1: Cohort 1:
  Placebo comparator is identical in appearance to the investigational product, containing the same excipients as the active comparator.
  The surgery for each subject is to be performed under general anesthesia supplemented by a transverse abdominis plane (TAP) block and local surgical site infiltration. Prior to the surgery, perform the TAP block as a single injection of 0.25% bupivacaine hydrochloride (HCl) 60 mL (150 mg).
  Placebo: Each cohort will use placebo reconstituted in saline.
  Bupivacaine Hydrochloride: 0.25% administered pre-surgery
  Hydromorphone: 0.02 mg/kg IV administered intraoperatively
  Fentanyl: 100 mcg IV administered intraoperatively
  Acetaminophen: 1000 mg IV administered intraoperatively
  Oxycodone: 5-10 mg PO administered post-surgery
- Placebo for Cohorts 2 and 3: Cohorts 2 & 3:
  Placebo comparator in each cohort is identical in appearance to the investigational product, containing the same excipients as the active comparator.
  The surgery for each subject is to be performed under general anesthesia supplemented by a transverse abdominis plane (TAP) block and local surgical site infiltration. Prior to the surgery, perform the TAP block as a single injection of 0.25% bupivacaine hydrochloride (HCl) 60 mL (150 mg).
  Placebo: Each cohort will use placebo reconstituted in saline.
  Bupivacaine Hydrochloride: 0.25% administered pre-surgery
  Hydromorphone: 0.02 mg/kg IV administered intraoperatively
  Fentanyl: 100 mcg IV administered intraoperatively
  Acetaminophen: 1000 mg IV administered intraoperatively
  Oxycodone: 5-10 mg PO administered post-surgery
Arm/Group | CA-008 5 mg (0.05 mg/mL) Cohort 1 | Placebo for Cohort 1 | CA-008 10 mg (0.1 mg/mL) | CA-008 15 mg (0.15 mg/mL) | Placebo for Cohorts 2 and 3
Number analyzed (Participants) | 9 | 9 | 12 | 12 | 12
score on a scale | 2.8 (2.59) | 2.0 (2.12) | 3.0 (2.22) | 2.8 (3.10) | 1.8 (1.96)
Statistical Analysis 1: Comparison: CA-008 15 mg (0.15 mg/mL) vs Placebo for Cohorts 2 and 3; Test type: Superiority; p = 0.2912, ANOVA

2. Secondary Outcome: Weighted Sum of Pain Intensity (SPI) Assessments = AUC of NRS Scores
Description: Pain intensity scores (using a Numeric Rating Scale of pain intensity from 0-10 where 0 is no pain and 10 is the worst pain imaginable) from 0 to T96 hours
Time Frame: 0 to 96 hours
Population: Safety population
Measure: Mean (Standard Deviation); unit: score on a scale*hours
Arm/Group | CA-008 5 mg (0.05 mg/mL) Cohort 1 | Placebo for Cohort 1 | CA-008 10 mg (0.1 mg/mL) | CA-008 15 mg (0.15 mg/mL) | Placebo for Cohorts 2 and 3
Number analyzed (Participants) | 9 | 9 | 12 | 12 | 12
score on a scale*hours | 392.98 (138.191) | 392.67 (163.025) | 384.94 (136.551) | 406.88 (220.821) | 356.23 (175.969)
Statistical Analysis 1: Comparison: CA-008 15 mg (0.15 mg/mL) vs Placebo for Cohorts 2 and 3; Test type: Superiority; p = 0.4980, ANOVA

3. Secondary Outcome: Time to Opioid Cessation or Freedom
Description: Time to the last use of opioid
Time Frame: From Surgery to Day 29
Population: Safety population
Measure: Median (Full Range); unit: hours
Arm/Group | CA-008 5 mg (0.05 mg/mL) Cohort 1 | Placebo for Cohort 1 | CA-008 10 mg (0.1 mg/mL) | CA-008 15 mg (0.15 mg/mL) | Placebo for Cohorts 2 and 3
Number analyzed (Participants) | 9 | 9 | 12 | 12 | 12
hours | 56.37 [1.25 to 216.65] | 55.42 [1.08 to 156.20] | 83.89 [0.95 to 323.22] | 59.55 [1.13 to 362.63] | 42.26 [1.02 to 238.57]
Statistical Analysis 1: Comparison: CA-008 15 mg (0.15 mg/mL) vs Placebo for Cohorts 2 and 3; Test type: Superiority; p = 0.1958, Log Rank

4. Secondary Outcome: Percent of Opioid Free Subjects
Description: Percent of subjects who were opioid free at 24-96 hours
Time Frame: 24 to 96 hours
Population: Safety population
Measure: Count of Participants; unit: Participants
Arm/Group | CA-008 5 mg (0.05 mg/mL) Cohort 1 | Placebo for Cohort 1 | CA-008 10 mg (0.1 mg/mL) | CA-008 15 mg (0.15 mg/mL) | Placebo for Cohorts 2 and 3
Number analyzed (Participants) | 9 | 9 | 12 | 12 | 12
Participants | 0 | 0 | 1 | 1 | 0
Statistical Analysis 1: Comparison: CA-008 15 mg (0.15 mg/mL) vs Placebo for Cohorts 2 and 3; Test type: Superiority; p = 0.9546, Regression, Logistic

5. Secondary Outcome: Total Opioid Consumption
Description: The sum of daily opioid consumption (in morphine equivalents)
Time Frame: 0 to 96 hours
Population: Safety population
Measure: Mean (Standard Deviation); unit: mg morphine equivalents
Arm/Group | CA-008 5 mg (0.05 mg/mL) Cohort 1 | Placebo for Cohort 1 | CA-008 10 mg (0.1 mg/mL) | CA-008 15 mg (0.15 mg/mL) | Placebo for Cohorts 2 and 3
Number analyzed (Participants) | 9 | 9 | 12 | 12 | 12
mg morphine equivalents | 85.83 (52.246) | 96.67 (63.134) | 69.77 (41.710) | 58.00 (69.170) | 77.85 (72.524)
Statistical Analysis 1: Comparison: CA-008 15 mg (0.15 mg/mL) vs Placebo for Cohorts 2 and 3; Test type: Superiority; p = 0.4434, ANOVA

ADVERSE EVENTS:
Time Frame: Approximately 76 days per subject from screening to the day 29 (D29) visit (however this could be longer to follow any AE to resolution or establishment of a new baseline)
Arm/Group | CA-008 5 mg (0.05 mg/mL) Cohort 1 | Placebo for Cohort 1 | CA-008 10 mg (0.1 mg/mL) | CA-008 15 mg (0.15 mg/mL) | Placebo for Cohorts 2 and 3
All-Cause Mortality (participants affected / at risk) | 0/9 | 0/9 | 0/12 | 0/12 | 0/12
Serious Adverse Events (participants affected / at risk) | 2/9 | 0/9 | 1/12 | 1/12 | 0/12
Other Adverse Events (participants affected / at risk) | 9/9 | 8/9 | 11/12 | 10/12 | 11/12
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | CA-008 5 mg (0.05 mg/mL) Cohort 1 (N=9) | Placebo for Cohort 1 (N=9) | CA-008 10 mg (0.1 mg/mL) (N=12) | CA-008 15 mg (0.15 mg/mL) (N=12) | Placebo for Cohorts 2 and 3 (N=12)
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Abortion spontaneous (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Deep vein thrombosis (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | CA-008 5 mg (0.05 mg/mL) Cohort 1 (N=9) | Placebo for Cohort 1 (N=9) | CA-008 10 mg (0.1 mg/mL) (N=12) | CA-008 15 mg (0.15 mg/mL) (N=12) | Placebo for Cohorts 2 and 3 (N=12)
Constipation (Gastrointestinal disorders) | 3 (3) | 2 (2) | 1 (1) | 2 (2) | 4 (4)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Lip oedema (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 5 (5) | 8 (8) | 6 (6) | 5 (5) | 3 (3)
Toothache (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0) | 2 (2) | 0 (0)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Incision site cellulitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Abdominal wound dehiscence (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Airway complication of anaesthesia (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Arthropod bite (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Flap necrosis (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Incision site pruritus (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Post procedural haematoma (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Seroma (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Wound dehiscence (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Transaminases increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 3 (3) | 4 (4) | 3 (3) | 4 (4) | 5 (5)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 4 (4) | 1 (1) | 1 (1) | 2 (2) | 2 (2)
Sciatica (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Abortion spontaneous (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Anxiety (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dermatitis contact (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Pruritus generalized (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Rash macular (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Deep vein thrombosis (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Phlebitis (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2019-01-28): https://cdn.clinicaltrials.gov/large-docs/18/NCT03789318/Prot_000.pdf
  • Statistical Analysis Plan (2019-04-24): https://cdn.clinicaltrials.gov/large-docs/18/NCT03789318/SAP_001.pdf